CLINICAL TRIAL: NCT03077321
Title: Improving Access to a Primary Care Based Positive Parenting Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 17-0545
Record Dates: First submitted 2017-03-02; First posted 2017-03-10 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Program Implementation; Child Behavior Problem; Positive Parenting

STUDY DESIGN:
Intervention Model Description: RCT 1:1:1
Who Masked: Investigator, Outcomes Assessor
Masking Description: The therapists and the parents will not be blinded to group because they will be providing and receiving the intervention. The investigators who are collecting the data will be blinded to arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CARE (Active Comparator): The parent-child dyads in the CARE arm will receive the standard CARE program.
  Interventions: Behavioral: CARE
- CARE plus peer mentor (Experimental): The parent-child dyads in the CARE plus peer mentor arm will receive the CARE program that is delivered with the peer mentor.
  Interventions: Behavioral: CARE plus Peer Mentor
- Control (No Intervention): Wait list control

INTERVENTIONS:
Behavioral: CARE plus Peer Mentor — A parent who has completed the standard CARE program will be recruited to be a peer mentor. The peer mentor will attend the CARE training for group leaders and will also be trained in motivational interviewing. These skills will then be used strategically in weekly phone discussions between the peer mentor and parent about practicing the CARE parenting skills in the home setting and planning for attending the 6 training sessions. The parent mentor will co-facilitate the CARE groups in the peer mentor arm along with 2 additional CARE therapists. The peer mentor will also call the parents in the peer mentor arm before each session to discuss progress on homework, and to address barriers for program attendance.
  Arms: CARE plus peer mentor
Behavioral: CARE — CARE involves 6 weekly 90-minute sessions administered to 6-10 parents by 2 therapists. The initial phase focuses on developing parenting skills aimed at increasing attention to children's pro-social behaviors while ignoring minor attention seeking misbehaviors. The second phase teaches techniques for giving children effective commands in order to set age-appropriate limits and increase compliance. Children do not attend the training but parents are expected to practice the skills with their children between sessions.
  Arms: CARE

SUMMARY:
This is a randomized clinical trial of the impact of incorporating a peer mentor into a primary care based group parenting program on increasing program participation by parents and improving program outcomes.

DETAILED DESCRIPTION:
The investigators will perform a randomized controlled trial of the impact of Child Adult Relationship Enhancement (CARE) plus peer mentor on increasing program adoption, acceptability, and appropriateness among 2-6 year old children and their parents at UNC Children's Primary Care Clinic. The investigators will also examine the effectiveness of CARE plus peer mentor on dysfunctional parenting and child behavior problems. Participants will be randomized to CARE plus peer mentor or standard CARE. Program attendance, acceptability, and appropriateness will be measured upon completion of the 6-week program. Dysfunctional parenting and child behavior will be measured at baseline and 6 weeks. The investigators will conduct semi-structured interviews among a sample of parents (~20-30) in order to understand the impact of the peer mentors on program implementation, as well as barriers and facilitators to program initiation and long-term participation.

ELIGIBILITY:
Inclusion Criteria:

* 2-6 year old child at UNC Children's Primary Care Clinic and their parent
* English speaking

Exclusion Criteria:

* child is developmentally younger than 2 years old
* child is already received mental health services for behavioral problems

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Program Adoption | 6-12 weeks
  mean number of sessions attended

SECONDARY OUTCOMES:
Child Behavior | 0 weeks and 6-12 weeks
  Child behavior as measured by the Eyberg Child Behavior Inventory. The Eyberg Child Behavior Inventory (ECBI) is a 36 item paper-and-pencil rating scales completed by parents that assesses the severity of conduct problems in children as well as the extent to which parents find the behaviors troublesome. It assesses the frequency of disruptive behaviors occurring in the home setting. It provides an Intensity Raw Score and a Problem Raw Score. The intensity scale (range 36-252) and the problem scale (range 0-36). In both cases higher values indicate more externalizing behaviors.
Dysfunctional Parenting Behaviors | 0 weeks and 6-12 weeks
  Dysfunctional parenting Behaviors as measured by the Parenting Scale.The Parenting Scale is a 30-item parent-report instrument that measures dysfunctional parenting practices for parents of young children. Specifically, the Parenting Scale measures laxness (permissive, inconsistent discipline); over-reactivity (harsh, emotional, authoritarian discipline); and hostility (use of verbal or physical force). It provides a total score, and three sub scale scores (laxness, over-reactivity, and hostility), each with a range of 1-7. Higher scores are indicative of more dysfunctional parenting.
Dysfunctional Parenting Attitudes | 0 weeks and 6-12 weeks
  Dysfunctional parenting attitudes as measured by the Adult Adolescent Parenting Inventory-2.The AAPI-2 is a 40 item self-report measure. The AAPI-2 assesses parenting attitudes along 5 dimensions: (1) inappropriate expectations of children, (2) parental lack of empathy towards children's needs, (3) strong belief in the use of corporal punishment as a means of discipline, (4) reversing parent-child role responsibilities, and (5) oppressing children's power and independence. Raw scores with a range from 1 to 10 are provided for each dimension and translated into risk categories: high (1-3), medium (4-7), low(8-10).

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Schilling, MD, MSHP, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to share the data with other researchers.

REFERENCES:
- [Derived] Schilling S, Ritter V, Wood JN, Fine J, Zolotor AJ. Child-Adult Relationship Enhancement in Primary Care: A Randomized Trial of a Skill-Based Parent Training with Parent Mentor Adaptation. J Dev Behav Pediatr. 2020 May;41(4):272-280. doi: 10.1097/DBP.0000000000000759. PMID 31809392